CLINICAL TRIAL: NCT02550353
Title: Comparison of Early Changes in Ocular Surface and Inflammatory Mediators Between Lenticule Extraction and Femtosecond Laser-assisted Laser in Situ Keratomileusis
Brief Title: Changes Between Lenticule Extraction and Femtosecond Laser-assisted Laser in Situ Keratomileusis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xingwu Zhong, MD PhD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-002
Record Dates: First submitted 2015-09-13; First posted 2015-09-15 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Myopia; Astigmatism
Keywords: lenticule extraction; femtosecond laser-assisted laser in situ keratomileusis; tear; inflammatory mediators
MeSH Terms: conditions — Myopia; Astigmatism; Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lenticule extraction (Experimental): The patients in this group chose to receive the lenticule extraction surgery
  Interventions: Procedure: lenticule extraction
- FS assisted laser in situ keratomileusis (Experimental): The patients in this group chose to receive the femtosecond laser-assisted laser in situ keratomileusis surgery.
  Interventions: Procedure: femtosecond laser-assisted laser in situ keratomileusis

INTERVENTIONS:
Procedure: lenticule extraction — Four femtosecond incisions were created in succession: the posterior surface of the refractive lenticule (spiral in), the lenticule border, the anterior surface of the refractive lenticule (spiral out), and the corneal flap in the superior region. After the suction was released, the flap was opened using a thin, blunt spatula and the free refractive lenticule was subsequently grasped with a forceps and extracted, after which the flap was repositioned carefully.
  Arms: lenticule extraction
Procedure: femtosecond laser-assisted laser in situ keratomileusis — track distance and spot distance were 3.0 μm during flap creation and 1.5 μm during flap side-cutting. The flap diameter was 8.0 mm, and flap thickness was set to 105 μm. Side-cut angle and hinge angle were 90°and 50° respectively. The flaps were created by laser scanning in spirals from the periphery to the center of the pupil. An excimer laser system was used in the subsequent ablation of the stromal bed with a 6.0 mm optical zone. Once the excimer ablation was completed, the flap was repositioned in a similar fashion as in routine LASIK.
  Arms: FS assisted laser in situ keratomileusis

SUMMARY:
The aim is to evaluate the short-term changes in ocular surface measures and tear inflammatory mediators after lenticule extraction (FLEx) and femtosecond laser-assisted laser in situ keratomileusis (FS-LASIK) procedures.

DETAILED DESCRIPTION:
Over the past few years, laser in situ keratomileusis with a femtosecond laser-created flap (FS-LASIK)has been a popular ophthalmic procedure for the correction of refractive error. This first all-in-one FS-laser system was designed to perform the refractive lenticule extraction (ReLEx) procedures, femtosecond lenticule extraction (FLEx).They have the same feature: corneal flap.

Ocular surface disruption during corneal refractive surgery is commonly considered to be closely related to the development of dry eye. Multiple etiologies contribute to this ocular surface disruption, including the flap creation and stromal ablation involved in previous refractive surgery techniques. Corneal nerve damage has been considered the main cause of dry eye, due to disrupted afferent sensory nerves, reduced blink reflex, and increased tear evaporation leading to tear film instability. In addition, postoperative inflammatory mediator fluctuations are also a key factor related to ocular surface damage. Extensive research has described the effects of cytokines, chemokines and growth factors in modulating corneal wound healing, cell migration, and apoptosis on the ocular surface after refractive surgery.

This prospective clinical study is going to assess the short-term changes in ocular surface measures and tear inflammatory mediators after lenticule extraction (FLEx) and femtosecond laser-assisted laser in situ keratomileusis (FS-LASIK) procedures.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years(range from 18 year to 25 years)
* corneal thickness 500 μm with calculated residual stromal bed after treatment greater than 300 μm
* preoperative spherical equivalent refraction between- 2.00 diopter (D) and -6.50 D.preoperative cylindrical equivalent refraction between -0.25 D and -1.50 D.
* preoperative corneal curvature from 41.0 D to 46.0 D with a regular topographic pattern monocular best corrected visual acuity of 20/20 or better and stable refractive error (less than 0.5 D change) for 24 months before surgery。

Exclusion Criteria:

* systemic disease that contraindicated the surgery (such as diabetes, glaucoma and systemic collagen vascular disease)
* corneal abnormality or disease.
* a history of tear supplement usage or contact lens wear during the past year.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Schirmer I test | up to 1month after surgery
corneal fluorescein staining | up to 1month after surgery
noninvasive tear breakup time | up to 1month after surgery
ocular surface disease index | up to 1month after surgery
central corneal sensitivity | up to 1month after surgery
tear meniscus height | up to 1month after surgery
Interleukin-1α | up to 1month after surgery
tumor necrosis factor-α | up to 1month after surgery
nerve growth factor | up to 1month after surgery
interferon-γ | up to 1month after surgery
transforming growth factor-β1 | up to 1month after surgery
matrix metalloproteinase-9 | up to 1month after surgery

SECONDARY OUTCOMES:
Correlation Between Inflammatory Mediators and Ocular Surface Changes | up to 1month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xingwu Zhong, MD,PhD, Principal Investigator — Hainan Eye Hospital, Zhongshan Ophthalmic Center of Sun Yat-sen University
Locations (1):
- Hainan Eye Hospital, Zhongshan Ophthalmic Center of Sun Yat-sen University, Haikou, Hainan, China